CLINICAL TRIAL: NCT02775500
Title: Apremilast Pregnancy Exposure Registry OTIS Autoimmune Diseases in Pregnancy Project
Brief Title: Apremilast Pregnancy Exposure Registry
Status: Active, not recruiting | Type: Observational
Sponsor: University of California, San Diego (Other)
Collaborators: Celgene (Industry); The Organization of Teratology Information Specialists (Other)
Responsible Party: Principal Investigator, Christina Chambers, Professor, Co-Director Center for Promotion of Maternal Health and Infant Development, University of California, San Diego
Other Study IDs: 141041
Record Dates: First submitted 2016-01-26; First posted 2016-05-17 (Estimated); Last update posted 2025-01-28 (Actual); Status verified 2025-01

CONDITIONS: Psoriatic Arthritis; Psoriasis
Keywords: pregnancy; apremilast; Otezla; autoimmune disease; psoriatic arthritis; psoriasis; TNF; tumor necrosis factor; birth outcome; birth defect
MeSH Terms: conditions — Arthritis, Psoriatic; Psoriasis; Autoimmune Diseases; Congenital Abnormalities | interventions — apremilast

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (4):
- Apremilast-Exposed Cohort: Women who have been exposed to apremilast in pregnancy for an approved indication in the first trimester of pregnancy for any length of time from the date of conception.
  Interventions: Drug: apremilast
- Diseased Comparison Cohort: Women with an approved disease who have not been exposed to apremilast at any time in pregnancy.
- Healthy Comparison Cohort: Healthy women who have no diagnosis of an approved indication or other chronic illness, have not taken apremilast in pregnancy, nor have they been exposed to any known human teratogen during pregnancy.
- Apremilast-Exposed Registry Group: Women who have been exposed to apremilast in pregnancy, for any length of time following the first day of the last menstrual period until the end of pregnancy who do not qualify for the prospective cohort study.
  Interventions: Drug: apremilast

INTERVENTIONS:
Drug: apremilast — Comparison of women exposed during pregnancy versus women who are not exposed to apremilast
  Other Names: Otezla
  Groups: Apremilast-Exposed Cohort; Apremilast-Exposed Registry Group

SUMMARY:
The purpose of the Apremilast Pregnancy Exposure Registry is to monitor planned and unplanned pregnancies exposed to apremilast and to evaluate the safety of this medication relative to specified pregnancy outcomes, and to evaluate potential effects of prenatal apremilast exposure on infant health status through one year of age.

DETAILED DESCRIPTION:
The Apremilast Pregnancy Exposure Registry (Registry) is a United States (U.S.) based registry designed to monitor planned or unplanned pregnancies exposed to apremilast when used to treat an approved indication in accordance with the current approved prescribing information, who reside in the U.S. or Canada.

The goal of the Registry is to conduct an observational, controlled prospective cohort study that will involve follow-up of live born infants to one year of age.

The primary objective of the Registry is to evaluate any potential increase in the risk of major birth defects, specifically a pattern of anomalies, in apremilast exposed pregnancies compared to the primary comparison group of disease-matched unexposed pregnancies. Secondary objectives are to evaluate the potential effect of exposure relative to the secondary comparison group of healthy pregnant women, and the effect of exposure on other adverse pregnancy outcomes including spontaneous abortion or stillbirth, preterm delivery, reduced infant birth size, a pattern of minor malformations, postnatal growth of live born children to one year of age, and incidence of serious or opportunistic infections or malignancies in live born children up to one year of age.

The Pregnancy Exposure Registry is sponsored by Celgene Corporation and is conducted by the Organization of Teratology Information Specialists (OTIS) Research Group and is administered by investigators at the coordinating site located at the University of California, San Diego. The study is planned for seven years.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant

Exclusion Criteria:

-

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The study population includes pregnant women who reside in the U.S. or Canada. All exposed subjects and comparison subjects will be recruited through spontaneous callers to participating OTIS member services in locations throughout North America and through active recruitment strategies, e.g., direct mailings to rheumatologists, dermatologists and other relevant specialists, obstetric health care providers, pharmacists, web site, and professional meetings.
Sampling Method: Non-Probability Sample
Enrollment: 233 (Actual)
Dates: Start 2014-11 (Actual); Primary Completion 2024-12 (Actual); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
The number of major structural malformations identified in the children of study participants | Throughout pregnancy through 1 year of life
  The primary objective of the study is to evaluate the effect of certain medications when used in the first trimester of pregnancy with respect to major structural birth defects in children of study participants. The study is analyzing the difference in the number of major malformations in children whose moms were exposed to apremilast compared to women without exposure to apremilast. Information will be collected from maternal interview and through medical records.
A pattern of major malformations identified in the children of study participants | Throughout pregnancy through 1 year of life
  The primary objective of the study is to evaluate the effect of certain medications when used in the first trimester of pregnancy with respect to a pattern of major malformations in children of study participants. The study is analyzing the difference in the pattern of major malformations in children whose moms were exposed to apremilast compared to women without exposure to apremilast. Information will be collected from maternal interview and through medical records.

SECONDARY OUTCOMES:
Pattern of minor structural malformations identified by study physical exam in the children of study participants | Assessed when the dysmorphology exam is conducted, which will occur between birth of the child and through study completion, an average of 1 year of age
  One secondary objective of the study is to evaluate the effects of certain medications when used in the first trimester of pregnancy with respect to a potential pattern of minor malformations. Information collected during the dysmorphology exam.
Pregnancy Outcome; rate of live born infants, spontaneous abortions, stillbirths, and terminations between cohort groups | At the end of pregnancy
  Another objective of the study is to evaluate the effects of certain medications when used in the first trimester of pregnancy with respect to pregnancy outcome (rates of live born infants, spontaneous abortions, stillbirths, and terminations. Information will be collected from maternal interview and through medical records.
Gestational age at delivery among infants in the cohort groups | At the end of pregnancy
  Another objective of the study is to evaluate the effects of certain medications when used in the first trimester of pregnancy with respect to gestational age at delivery. Rates of preterm and full-term delivery between cohorts will be compared, as well as any statistical differences in gestational age at delivery. Information will be collected from maternal interview and through medical records.
Pregnancy Complication rates between cohort groups | From the first day of the last menstrual period (LMP) through delivery
  Another objective of the study is to evaluate the effects of certain medications when used in the first trimester of pregnancy with respect to pregnancy complications. Rates of pregnancy complications between cohorts will be compared. Information will be collected from maternal interview and through medical records.
Neonatal Complication rates between cohort groups | Birth of the child to 1 month of age.
  Another objective of the study is to evaluate the effects of certain medications when used in the first trimester of pregnancy with respect to neonatal complications. Rates of neonatal complications between cohorts will be compared. Information will be collected from maternal interview and through medical records.
Pre- and post-natal fetal and infant growth percentiles | From the first day of the last menstrual period (LMP) through delivery, and up to one year of age of the child
  Pre- and post-natal fetal and infant growth will be compared between cohorts. The study will analyze rates between cohorts for small for gestational age, those that are small for weight, length, and/or head circumference up to one year of age. Information will be collected from maternal interview and through medical records.
Any serious and opportunistic infections rates occurring in infants whose mothers are enrolled in the study | Up to one year of age of the child
  Any opportunistic or serious infection, including any infection requiring hospitalization in the child. Rates of infections will be compared between cohort groups. Information will be collected from maternal interview and through medical records.
Any malignancies diagnosed in infants of mothers enrolled in the study | Up to one year of age of the child
  Any malignancy diagnosed in the child up to 1 year of age. Rate of malignancies will be compared between cohort groups. Information will be collected from maternal interview and through medical records.

CONTACTS AND LOCATIONS:
Overall Officials: Christina Chambers, PhD, MPH, Principal Investigator — UCSD
Locations (1):
- University of California, San Diego, La Jolla, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Organization of Teratology Information Specialists and MotherToBaby website containing study information — https://mothertobaby.org/pregnancy-studies/